CLINICAL TRIAL: NCT07158307
Title: Safety and Efficacy of Paclitaxel-coated PTCA Balloon Catheter With a Shellac Plus Vitamin E Excipient (GENOSS® DCB) in Patients With De Novo Lesion of Small Coronary Artery Disease: A Prospective, Multi-center, Observational Study
Brief Title: Safety and Efficacy of GENOSS® DCB With a Shellac Plus Vitamin E Excipient in Patients With De Novo Lesion
Acronym: PCB-De Novo
Status: Enrolling by invitation | Type: Observational
Sponsor: Genoss Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP-DS1001-3
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease(CAD)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- GENOSS® DCB (Paclitaxel-coated PTCA Balloon Catheter): Patients with de novo small coronary artery disease who underwent PCI with GENOSS DCB

SUMMARY:
The GENOSS PCB-De Novo study aims to evaluate the long-term efficacy and safety of a paclitaxel-coated balloon catheter containing shellac and vitamin E excipients (Genoss® DCB) in patients with De novo small coronary artery disease.

DETAILED DESCRIPTION:
This prospective, open-label, multicenter, observational study will enroll patients with de novo small coronary artery disease undergoing PCI with the GENOSS® DCB at 47 hospitals.

Because this is an observational study, the number of participants will not be calculated separately, but a total of 3,000 participants are planned to be recruited during the study enrollment period.

All patients will be followed up at 1, 2, and 3 years postprocedure to evaluate the safety and efficacy of the paclitaxel-coated PTCA balloon catheter.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 19
* Patients with new lesions with coronary small vascular disease (vascular diameter <3.0 mm) underwent a GENOSS® DCB procedure through percutaneous coronary intervention
* Subjects who agreed to the clinical research plan and the clinical follow-up plan, voluntarily decided to participate in this clinical study, and agreed in writing to the consent of the study subjects

Exclusion Criteria:

* Subjects who plan to become pregnant during the period of this study as women of the gestational age
* Subjects whose remaining life expectancy is expected to be less than one year
* Subjects who visited the hospital due to psychogenic shock at the time of visiting the hospital and are predicted to have a low chance of survival based on medical judgment
* If it falls under any of the following items after prior dilation of the target lesion;

  * Stent procedures are required due to vascular detachment that limits blood flow
  * If the residual stenosis is >30%
  * If the TIMI flow is <3
* Subjects participating in a randomized study of medical devices
* If the researcher determines that it is not appropriate for this clinical study or may increase the risk associated with participation in the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who underwent PCI with GENOSS DCB for small coronary artery disease with de novo lesions
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2030-06-27 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Target lesion failure (TLF) | at 1 year after the procedure
  composite endpoint of cardiac death, target vessel myocardial infarction, and ischemia-driven target lesion revascularization

SECONDARY OUTCOMES:
Target lesion failure (TLF) | at 2, 3 years after the procedure
  composite endpoint of cardiac death, target vessel myocardial infarction, and ischemia-driven target lesion revascularization
Major cardiac adverse events (MACE) | at 1, 2, 3 years after the procedure
  composite endpoint of death, myocardial infarction, and revascularization
all mortality | at 1, 2, 3 years after the procedure
  all deaths and cardiac deaths
any MI | at 1, 2, 3 years after the procedure
  all myocardial infarction and target vessel myocardial infarction (TV-MI)
all revascularization and ischemia-driven target lesion revascularization (ID-TLR) | at 1, 2, 3 years after the procedure
major bleeding event | at 1, 2, 3 years after the procedure
  BARC 3, 5

CONTACTS AND LOCATIONS:
Locations (1):
- Ulsan University Hospital, Ulsan, South Korea

IPD SHARING:
Plan to Share IPD: No